CLINICAL TRIAL: NCT02273362
Title: Pilot Study of EGFR Inhibition With Erlotinib in Cirrhosis to Inhibit Fibrogenesis and Prevent Hepatocellular Carcinoma
Brief Title: Erlotinib Hydrochloride in Preventing Liver Cancer in Patients With Cirrhosis of the Liver
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2014-02170; NCI-2014-02170 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HHSN261201200042I; N01-CN-2012-00042; MAY2013-02-02 (Other: Mayo Clinic in Rochester); MAY2013-02-02 (Other: DCP); N01CN00042 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2022-02-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Cirrhosis; Hepatocellular Carcinoma
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevention (erlotinib hydrochloride) (Experimental): Patients receive erlotinib hydrochloride PO QD for 7 days (depending on the date of surgery, treatment range may be 5-14 days).
  Interventions: Drug: Erlotinib; Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Erlotinib — Given PO
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot phase I/II trial studies the best dose of erlotinib hydrochloride and to see how well it works in preventing liver cancer in patients with scarring (cirrhosis) of the liver. Erlotinib hydrochloride may help to inhibit the development of fibrous tissue and prevent liver cancer from forming in patients with cirrhosis of the liver.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safe and minimum effective dose (MED) of daily erlotinib (erlotinib hydrochloride) that inhibits epidermal growth factor receptor (EGFR) signaling in the target organ (liver) as assessed by phosphorylated (phospho)-EGFR staining.

SECONDARY OBJECTIVES:

I. Determine the relationship between erlotinib dose-schedule and side effects in participants with cirrhosis.

TRANSLATIONAL OBJECTIVES:

I. Determine the relationship between erlotinib dose-schedule and immuno-histochemical staining pattern of phospho-ERK, proliferating cell nuclear antigen (PCNA), epidermal growth factor (EGF), and alpha smooth muscle actin (alphaSMA) in the liver.

II. Determine the relationship between erlotinib dose-schedule and gene expression signature associated with prognosis in cirrhosis participants following hepatocellular carcinoma (HCC) resection.

III. Determine the relationship between erlotinib dose-schedule and viral load in participants with hepatitis C virus (HCV) positive (+).

IV. Determine the relationship between erlotinib dose-schedule and erlotinib plasma level on day of liver resection.

OUTLINE: This is a phase I, dose-escalation/de-escalation study followed by a phase II study.

Patients receive erlotinib hydrochloride orally (PO) once daily (QD) for 7 days (depending on the date of surgery, treatment range may be 5-14 days).

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION:
* Individuals with a clinical diagnosis fibrosis or cirrhosis of the liver (no more than Child-Pugh classification A; Child-Pugh-Turcotte score of 6 or less) who have:

  * An indication for surgical liver resection, OR
  * A clinical liver biopsy (with research tissue specimens available for analysis) =< 3 months prior to pre-registration
* Willingness to discontinue smoking during the study two weeks prior to beginning the study and willingness to not smoke while taking study medication
* Not pregnant or breast feeding. Note: The effects of erlotinib (Tarceva) on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.
* Willingness to use adequate contraception to avoid pregnancy or impregnation until 2 weeks after discontinuing study agent
* Willingness to provide mandatory blood specimens
* Able to undergo:

  * Percutaneous or transjugular biopsy of cirrhotic liver at least 7 days prior to liver resection (surgical cohort), OR
  * A biopsy of the cirrhotic liver (non-surgical cohort)
* Willingness to authorize collection of tissue from surgically-resected liver or clinical liver biopsy for analyses
* Ability to understand and the willingness to sign a written informed consent document
* REGISTRATION INCLUSION:
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* International normalized ratio (INR) =< 1.5
* Platelets >= 50 B/L (10^9/L)
* Total bilirubin =< 3 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x institutional ULN
* Creatinine =< 1.5 x institutional ULN
* Non-surgical cohort only: positive phospho-EGFR assessment (>= 100 stained pixels) from tissue obtained from previous clinical liver biopsy
* Pre-intervention biopsy sample collected

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION:
* Any prior treatment with erlotinib or other agent whose primary mechanism of action is known to inhibit EGFR
* Participants with a known diagnosis of human immunodeficiency virus (HIV); Note: an HIV screening test does not have to be performed to evaluate this criterion
* Participants who regularly (>= 2 times per week) use drugs that alter the pH of the gastrointestinal (GI) tract, such as proton pump inhibitors (PPI) and antacids; exceptions: individuals who use prescription PPIs and have approval from their primary health care provider to discontinue for the duration of clinical trial participation may be enrolled; an alternate drug to control gastroesophageal reflux disease (GERD)/peptic ulcer disease (PUD) symptoms will be suggested
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Use of potent CYP3A4 inhibitors, such as ketoconazole, atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole, and grapefruit or grapefruit juice
* Use of CYP3A4 inducers such as rifampicin, rifabutin, rifapentine, phenytoin, carbamazepine, phenobarbital, and St. John's wort
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib (Tarceva)
* Participants who cannot have their warfarin, Lovenox, Plavix, or other comparable medications held for percutaneous or transjugular liver biopsy and surgery if so indicated
* Non-surgical cohort only: pathology report from clinical liver biopsy (=< 3 months prior to pre-registration) demonstrates no histologic abnormalities associated with chronic hepatitis, steatohepatitis, fibrosis, or cirrhosis
* REGISTRATION EXCLUSION:
* Receiving any other investigational agents =< 6 months prior to registration
* Surgical cohort (cohort A only): percutaneous or transjugular biopsy incomplete or not performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K Tanabe, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mount Sinai Hospital, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Derived] Tanabe KK, Zahrieh D, Strand CA, Hoshida Y, Flotte TJ, Della'Zanna G, Umar A, Chavin KD, Cleary S, Kubota N, Llovet JM, Patel T, Siegel C, Limburg PJ. Epidermal Growth Factor Receptor Inhibition With Erlotinib in Liver: Dose De-Escalation Pilot Trial as an Initial Step in a Chemoprevention Strategy. Gastro Hep Adv. 2024 Jan 29;3(3):426-439. doi: 10.1016/j.gastha.2024.01.009. eCollection 2024. PMID 39131140

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 0 ( 75 mg Erlotinib Hydrochloride Daily): Patients receive 75 mg erlotinib hydrochloride PO QD for 7 days.
- Dose Level -1 (50 mg Erlotinib Daily): Patients receive 50 mg erlotinib hydrochloride PO QD for 7 days.
- Dose Level -2 (25 mg Erlotinib Daily): Patients receive 25 mg erlotinib hydrochloride PO QD for 7 days.
Period: Overall Study
Arm/Group | Dose Level 0 ( 75 mg Erlotinib Hydrochloride Daily) | Dose Level -1 (50 mg Erlotinib Daily) | Dose Level -2 (25 mg Erlotinib Daily)
Started | 5 | 6 | 14
Completed | 5 | 6 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients registered and treated per protocol are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 0 ( 75 mg Erlotinib Hydrochloride Daily) | Dose Level -1 (50 mg Erlotinib Daily) | Dose Level -2 (25 mg Erlotinib Daily) | Total
Number analyzed (Participants) | 5 | 6 | 14 | 25
Age, Continuous [Median (Full Range); unit: years] | 61 [55 to 76] | 58.5 [48 to 80] | 66 [38 to 75] | 64 [38 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 8
  Male | 3 | 4 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 3 | 4 | 11 | 18
  Unknown or Not Reported | 1 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 2 | 6 | 12 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Response (at Least a 50% Reduction in Liver Phospho-EGFR Staining)
Description: A response is defined as having at least a 50% reduction in liver phospho-EGFR staining (50% reduction in the percentage of positive pixels).> > For each dose level, we report the number of participants achieving a response (at least 50% reduction in liver phospho-EGFR staining). >
  > The Minimum effective dose (MED) is defined as the dose which at least a 40% of patients report a response.
Time Frame: Up to day 7
Population: In Dose Level 0, 1 participant terminated intervention early due to physician decision and 1 participant lost pre-intervention tissue specimens. 1 participant in dose level -1 terminated intervention early due to adverse event. In Dose Level -2, 3 participants did not have additional pre-intervention tissue specimens available beyond eligibility and 1 participant was not evaluable for phospho-EGFR staining at post-intervention due to no benign liver tissue.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0 ( 75 mg Erlotinib Hydrochloride Daily) | Dose Level -1 (50 mg Erlotinib Daily) | Dose Level -2 (25 mg Erlotinib Daily)
Number analyzed (Participants) | 3 | 5 | 10
Participants | 3 | 3 | 6

2. Secondary Outcome: Adverse Event Profile
Description: Graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4. For this endpoint, we are reporting the number of participants with Grade 3 or higher as their worst reported adverse event.
Time Frame: Up to day 7
Population: All patients that began protocol treatment are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0 ( 75 mg Erlotinib Hydrochloride Daily) | Dose Level -1 (50 mg Erlotinib Daily) | Dose Level -2 (25 mg Erlotinib Daily)
Number analyzed (Participants) | 5 | 6 | 14
Participants | 0 | 1 | 2

3. Other Pre Specified Outcome: Changes in Phospho-ERK Levels in the Liver
Description: The relationship between dose-level and staining of biomarkers in the liver will be assessed. The baseline biomarker expression levels across all the dose levels using analysis of variance (ANOVA) or the nonparametric equivalent will be compared. The changes in these biomarker values will be assessed using the Wilcoxon signed-rank test and compare these changes across dose levels using ANOVA. Graphical methods will be used to assess the differences in these biomarker values across dose levels. All categorical variables will be analyzed using chi-square or Fisher's exact tests.
Time Frame: Baseline to day 7
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Changes in PCNA Levels in the Liver
Description: The relationship between dose-level and staining of biomarkers in the liver will be assessed. The baseline biomarker expression levels across all the dose levels using ANOVA or the nonparametric equivalent will be compared. The changes in these biomarker values will be assessed using the Wilcoxon signed-rank test and compare these changes across dose levels using ANOVA. Graphical methods will be used to assess the differences in these biomarker values across dose levels. All categorical variables will be analyzed using chi-square or Fisher's exact tests.
Time Frame: Baseline to day 7
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Changes in EGF Levels in the Liver
Description: as for outcome 4
Time Frame: Baseline to day 7
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in alphaSMA Levels in the Liver
Description: as for outcome 4
Time Frame: Baseline to day 7
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Modulation of Gene Expression Signatures Associated With Prognosis in Cirrhosis
Description: The relationship between dose and modulation of a gene expression signature associated with prognosis in cirrhosis will be assessed. The baseline biomarker expression levels across all the dose levels using ANOVA or the nonparametric equivalent will be compared. The changes in these biomarker values will be assessed using the Wilcoxon signed-rank test and compare these changes across dose levels using ANOVA. Graphical methods will be used to assess the differences in these biomarker values across dose levels. All categorical variables will be analyzed using chi-square or Fisher's exact tests.
Time Frame: Baseline to day 7
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Viral Load in Participants With Hepatitis C Virus (HCV)+
Description: Whether erlotinib hydrochloride is associated with a measurable reduction in viral load in participants with HCV+ will be determined. The baseline biomarker expression levels across all the dose levels using ANOVA or the nonparametric equivalent will be compared. The changes in these biomarker values will be assessed using the Wilcoxon signed-rank test and compare these changes across dose levels using ANOVA. Graphical methods will be used to assess the differences in these biomarker values across dose levels. All categorical variables will be analyzed using chi-square or Fisher's exact tests.
Time Frame: Baseline to 7 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Erlotinib Hydrochloride Plasma Level
Description: The relationship between erlotinib hydrochloride dose-schedule and erlotinib hydrochloride plasma level on the day of liver resection will be determined.
Time Frame: Day of liver resection
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Dose Level 0 ( 75 mg Erlotinib Hydrochloride Daily) | Dose Level -1 (50 mg Erlotinib Daily) | Dose Level -2 (25 mg Erlotinib Daily)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 1/14
Other Adverse Events (participants affected / at risk) | 2/5 | 4/6 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 ( 75 mg Erlotinib Hydrochloride Daily) (N=5) | Dose Level -1 (50 mg Erlotinib Daily) (N=6) | Dose Level -2 (25 mg Erlotinib Daily) (N=14)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 ( 75 mg Erlotinib Hydrochloride Daily) (N=5) | Dose Level -1 (50 mg Erlotinib Daily) (N=6) | Dose Level -2 (25 mg Erlotinib Daily) (N=14)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT02273362/Prot_SAP_000.pdf